CLINICAL TRIAL: NCT04911348
Title: Neurosarcoidosis : Initial Presentation and Disease Course, a Multicenter Retrospective Study
Brief Title: Neurosarcoidosis : Initial Presentation and Disease Course
Acronym: NEUROSARC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI207
Record Dates: First submitted 2021-02-18; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-02

CONDITIONS: Neurosarcoidosis
MeSH Terms: conditions — Neurosarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: none (observational) — no intervention

SUMMARY:
Neurosarcoidosis represents up to 10% of sarcoidosis cases. Little is known about its long-term course, even if the disease remains mainly monophasic with/w.o. sequelae, or if bouts of new symptoms may arise over years (polyphasic).

Using retrospective data from patients diagnosed with neurosarcoidosis in three French referral centers for neuro-inflammation, the investigators aim to determine patterns of disease course, according to the initial presentation and the treatments used.

DETAILED DESCRIPTION:
Sarcoidosis is a systemic inflammatory disease which a 10-20/100.000/year incidence rate. The nervous system is found to be affected in 5-10% in clinical series, rising to 14-27% in post-mortem studies. Mortality is as high as 5% mainly due to cardiac, pulmonary or neurological injury. The treatment of the disease uses cortico-steroids, and often steroid-sparing immunosuppressive agents such as methotrexate or cyclophosphamide. More recently, TNFalpha-blockers have been found to be highly effective.

Long-term data about the clinical and paraclinical course of the disease are lacking. "Bouts" or "relapse" of the disease are barely described, with no substantial information about their frequency, their sequelae, or their response to the treatments when initiated. Less is known about the risk of recurrence in each presentation of neurosarcoidosis (peripheral, spinal, brain or meningeal presentations). In the end, if a truly relapsing-remitting form of the disease exist is not sure, many patients presenting with a lond-standing pattern of invariant symptoms.

Due to this lack of knowledge about the natural history of neurosarcoidosis, even a "good treatment response" cannot be defined, and in many cases, it is difficult to attribute to treatments a seemingly favourable course af the disease.

In the current study, the investigators aim to build a retrospective cohort of patients diagnosed with neurosarcoidosis and seen at least once in three French referral centers for neuro--inflammation from Jan-1st-2000 to date : Nancy (Lorraine, North-Eastern), Bordeaux (Aquitaine, South-Western) and Strasbourg (Alsace, North-Eastern).

Demographics, clinical and paraclinical data at presentation will be collected(magnetic resonance imaging of the spine and brain, electroneuromyography if available, data of blood and cerebro-spinal fluid). After having clustered patients by presentation pattern, data about lines and types of treatments, change in clinical and paraclinical data will be collected. From this perspective, patterns of disease course on the mid/long-term will be established.

Estimated number of patients : 60-100. Estimated duration of follow-up : 5-10 years. Intervention : none (existing data).

ELIGIBILITY:
Inclusion Criteria:

* To have at least one documented visit in one of the three referral neurological centers (Nancy, Bordeaux, Strasbourg) between Jan-1st-2000 and Jan-1st-2021
* To be diagnosed with possible/probable/definite neurosarcoidosis

Exclusion Criteria:

- Denial to participate to the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every patient of the three centers meeting the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
change in disease characteristics from Baseline to end of study | from baseline to end of study (an average of 6 years)
  composite variable with three categories : monophasic course / polyphasic course with the same symptoms / polyphasic course with different symptoms
  This variable is composite and its evaluated by the investigators by reviewing the medical file with every available document : MRI results, clinical evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Guillaume Mathey, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No